CLINICAL TRIAL: NCT04552080
Title: The Effect of Systemic Antibiotics on Post-surgical Complications and Patient-centered Outcomes in Patients Undergoing Implant Surgery With Guided Bone Regeneration and Simultaneous Sinus Floor Elevation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Syst AB + Sinus 01
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Patients Undergoing Oral Implant Therapy
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Amoxicillin (Active Comparator)
  Interventions: Drug: Amoxicillin
- Comparator: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Preoperatively antibiotics of 2 g amoxicillin 1 hour prior to standard implant placement and sinus floor Elevation will be administered. An additional single dose of 500 mg of amoxicillin will be administered 8 hours after surgery and 500 mg thrice daily (8 hourly) on days 1 to 3 following implant placement and sinus floor elevation.
  Arms: Test: Amoxicillin
Other: Placebo — Preoperatively a placebo of 2 g will be administered. An additional single dose of 500 mg of placebo will be administered 8 hours after surgery and 500 mg thrice daily (8 hourly) on days 1 to 3 following implant placement and sinus floor elevation.
  Arms: Comparator: Placebo

SUMMARY:
The primary aim of the trial is to evaluate the effect of systemic antibiotic administration compared to placebo in patients undergoing oral implant therapy with simultaneous lateral sinus floor elevation and guided bone regeneration (GBR) in regard to patient-centered outcomes.

The secondary aims of the trial is to evaluate the effect of systemic antibiotic administration on postsurgical complications, in patients undergoing oral implant therapy with simultaneous lateral approach sinus floor elevation and guided bone regeneration (GBR).

ELIGIBILITY:
Inclusion Criteria:

1. Medically healthy adult: ASA (American Society of Anesthesiologists) classification I-II, age ≥ 21 years old
2. Non-smoker, previous smoker (quit ≥ 5 years); light smoker with less than 10 cigarettes/ day
3. Not allergic to Amoxicillin/Penicillin antibiotics, NSAIDS (Nonsteroidal anti-inflammatory drugs) or corn-starch
4. Edentulous spaces in the posterior maxilla in one or 2 posterior quadrants with an alveolar bone defect requiring sinus floor elevation and allowing implant placement of up to 3 dental implants and simultaneous GBR (residual crest height 3-5 mm; per implant site (Felice et al. 2012; Park et al. 2019).
5. Absence of signs of pathology of the sinus membrane and acute sinusitis requiring ongoing management -

Exclusion Criteria:

1. Medically compromised subjects (ASA classification III-V)
2. General contraindications against implant treatment or augmentative procedures (e.g. immunodeficiency, advanced systemic diseases, corticosteroid medication)
3. Those taking Bisphosphonates/anti-angiogenic/RANKL (Receptor activator of nuclear factor kappa-Β Ligand) inhibitor medications or receiving local radio-therapy
4. Heavy smoker or previous heavy smoker (quit < 5 years; ≥ 10 cigarettes/day)
5. Allergic to Amoxicillin or Penicillin antibiotics, NSAIDS and / or corn starch
6. Use of any form of antibiotics in the last 3 months or subjects requiring regular antibiotic prophylaxis prior to dental treatment
7. Pregnant or breast feeding. Self-declared intend to conceive (A pregnancy test will be performed for all female patients).
8. Need for 2 stage sinus augmentation
9. Acute or unmanaged symptomatic sinusitis
10. Type 1 implant placement (immediate implant placement following extraction)
11. Need for simultaneous soft tissue augmentation
12. Residual bone height of > 5mm.
13. Subjects aged < 21 years old

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient-centered Outcomes - 1 | days 1-7 and 14
  Change in visual analogue scores (VAS) on the wound (pain, swelling, bruising, haematoma, bleeding) Intensity of bleeding, swelling, pain and bruising on a score from 1(mild) to 10(severe).
Patient-centered Outcomes - 2 | days 1-7 and 14
  Change in discomfort of the sinuses (nosebleed, nasal congestion, rhinorrhea, feeling of pressure, hyposmia)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, University Hospital for Dentistry and Oral Health, Graz, Austria

IPD SHARING:
Plan to Share IPD: No